CLINICAL TRIAL: NCT03639701
Title: Deoxythymidine and Deoxycytidine Treatment for Thymidine Kinase 2 (TK2) Deficiency
Brief Title: Treatment of TK2 Deficiency With Thymidine and Deoxycytidine
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Muscular Dystrophy Association (Other); Hospital Universitario 12 de Octubre (Other); Instituto de Salud Carlos III (Other Government); University of Seville (Other); Medical Research Council Mitochondrial Biology Unit (Unknown); Centro de Investigación Biomédica en Red Enfermedades Raras (CIBERER), Spain (Unknown); Hospitales Universitarios Virgen del Rocío (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ7552
Record Dates: First submitted 2018-08-07; First posted 2018-08-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial DNA Depletion Syndrome 2 Myopathic Type; Thymidine Kinase 2 Deficiency
Keywords: Thymidine; Deoxycytidine
MeSH Terms: interventions — Thymidine; Deoxycytidine

STUDY DESIGN:
Intervention Model Description: Open label treatment with thymidine and deoxycytidine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label thymidine and deoxycytidine (Experimental): All patients will receive open label thymidine and deoxycytidine
  Interventions: Drug: Thymidine

INTERVENTIONS:
Drug: Thymidine — Mitochondrial DNA nucleotide precursors. Dose escalation: 130mg/kg/day x 14 days, 260 mg/kg/day x 14 days, and 400mg/kg/day as tolerated. Compounds are taken orally and divided into 3 doses daily.
  Other Names: Deoxycytidine

SUMMARY:
Patients with confirmed mitochondrial DNA depletion syndrome 2 (thymidine kinase 2 [TK2] deficiency) have reduced levels of nucleotides (deoxythymidine monophosphate and deoxycytidine monophosphate) for mitochondrial DNA synthesis. This results in mitochondrial DNA depletion syndrome (i.e less number of functional mitochondrial DNA). Patients with confirmed TK2 deficiency will be treated with open label deoxythymidine (dThd) and deoxycytidine (dCyt), which are nucleotide precursors, with the expectation that the cells could make additional mitochondrial DNA. This in turn may help reduce the clinical symptoms.

DETAILED DESCRIPTION:
Mitochondrial are responsible for the production of cellular energy. Mitochondria contain DNA which is the encoding system ( "recipe") for making the proteins that allow the mitochondria to function. Reduced amount of mitochondrial DNA, caused by genetic mutations in certain genes, Mitochondrial DNA Depletion Syndrome. This can result in symptoms; such as fatigue, weakness, and deficiencies in various body systems. TK2 deficiency is considered a mitochondrial depletion syndrome. Patients with TK2 deficiency have weakness and walking difficulty. They also have depleted levels of chemicals (phosphorylated deoxythymidine and deoxycytidine) used to make mitochondrial DNA. Based on previous studies with a similar compound, patients reported more energy and better motor skills.

Eligible patients include those with genetic mutations in the TK2 gene who are willing to attend several outpatient visits, and have motor skills testing, neurological exam by doctor, and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of TK2 deficiency
* Deemed by principle investigator to be symptomatic with TK2 deficiency
* Single gene disease; absence of polygenic disease
* Hematocrit within normal range for age group
* Patient or patient's guardian able to consent and comply with protocol requirements
* Presence of caregiver to ensure study compliance (if needed)
* Abstention from use of all pill-form dietary supplements and non-prescribed medications (except as allowed by the investigator)
* Abstention from use of other investigational medications or other medications according to the study investigator

Exclusion Criteria:

* Clinical history of bleeding or abnormal prothrombin time (PT)/partial thromboplastin time (PTT)
* Hepatic insufficiency with liver function tests (LFTs) greater than two times normal
* Renal insufficiency requiring dialysis
* Any other concurrent inborn errors of metabolism
* Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase | Up to 60 months
  Number of participants with treatment-related elevated alanine aminotransferase (ALT) serum level relative to upper limit of normal (expressed as ratios) grade 3 or higher as defined by CTCAE 4.03.
Aspartate aminotransferase | Up to 60 months
  Number of participants with treatment-related elevated aspartate aminotransferase (AST) serum level relative to upper limit of normal (expressed as ratios) grade 3 or higher as defined by CTCAE 4.03.
Gamma-glutamyltransferase | Up to 60 months
  Number of participants with treatment-related elevated gamma-glutamyltransferase (GGT) serum level relative to upper limit of normal (expressed as ratios) grade 3 or higher as defined by CTCAE 4.03.
Blood lymphocyte count | Up to 60 months
  Blood lymphocyte count increased relative to upper limit or normal or decreased relative to lower limit of normal (expressed as ratios) grade 3 or higher as defined by CTCAE 4.03.
Creatinine | Up to 60 months
  Serum creatinine level increased relative to upper limit of normal (expressed as ratios) grade 3 or higher as defined by CTCAE 4.03.
Electrocardiogram | Up to 60 months
  Number of patients with treatment related electrocardiogram (ECG) QT corrected interval (QTc) grade 3 or higher as defined by CTCAE version 4.03.
Diarrhea | Up to 60 months
  Patient-Reported Outcome Measurement Information System (PROMIS) Scale v1.0 - Gastrointestinal Diarrhea 6a score (score range 0-30 with higher scores indicating more severe diarrhea)

SECONDARY OUTCOMES:
Event-free survival | Up to 60 months
  Time to mechanical ventilation, death, or both will be assessed.
6-minute walk test | Up to 60 months
  Distance walked in meters over 6 minutes will be measured in ambulatory patient.
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) | Up to 60 months
  Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) score (0-64 point range with higher scores indicating better function) will be assessed in infants to assess motor function.
Hammersmith Functional Motor Scale Expanded (HFMSE) | Up to 60 months
  Hammersmith Functional Motor Scale Expanded (HFMSE) score (0-66 point range with higher scores indicating better function) will be measured in subjects >1 year-old.
Vital Capacity | Up to 60 months
  Vital capacity (percent of predicted normal based on age and height) will be measure by spirometry
Time on Mechanical Ventilation | Up to 60 months
  Number of hours per day that subjects use mechanical ventilation will be recorded.
euro Quality of Life (Neuro-QoL) in adults | Up to 60 months
  Neuro Quality of Life (Neuro-QoL) short forms will be used to assess effects of muscle weakness on motor function and activities of daily living. In adults, Lower and Upper Extremity scales will be assessed (0-80 points with higher scores indicating better function).
Neuro Quality of Life (Neuro-QoL) in pediatric subjects | Up to 60 months
  Neuro Quality of Life (Neuro-QoL) forms will be used to assess effects of muscle weakness on motor function and activities of daily living. In pediatric subjects (<18 years-old), Lower and Upper Extremity scales will be assessed (0-160 points with higher scores indicating better function).
Suicidal Ideation | Up to 60 months
  Suicidal ideation will be assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS), which contains 6 "yes" or "no" questions. Answer of "yes" to any question indicates possible suicide risk and answer of "yes: to questions 4, 5, or 6 indicates high-risk.

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Since there are very few patients in the world with TK2 Deficiency, we may share de-identified data with other researchers who are treating patients with TK2 Deficiency

REFERENCES:
- [Result] Garone C, Taylor RW, Nascimento A, Poulton J, Fratter C, Dominguez-Gonzalez C, Evans JC, Loos M, Isohanni P, Suomalainen A, Ram D, Hughes MI, McFarland R, Barca E, Lopez Gomez C, Jayawant S, Thomas ND, Manzur AY, Kleinsteuber K, Martin MA, Kerr T, Gorman GS, Sommerville EW, Chinnery PF, Hofer M, Karch C, Ralph J, Camara Y, Madruga-Garrido M, Dominguez-Carral J, Ortez C, Emperador S, Montoya J, Chakrapani A, Kriger JF, Schoenaker R, Levin B, Thompson JLP, Long Y, Rahman S, Donati MA, DiMauro S, Hirano M. Retrospective natural history of thymidine kinase 2 deficiency. J Med Genet. 2018 Aug;55(8):515-521. doi: 10.1136/jmedgenet-2017-105012. Epub 2018 Mar 30. PMID 29602790
- [Result] Lopez-Gomez C, Levy RJ, Sanchez-Quintero MJ, Juanola-Falgarona M, Barca E, Garcia-Diaz B, Tadesse S, Garone C, Hirano M. Deoxycytidine and Deoxythymidine Treatment for Thymidine Kinase 2 Deficiency. Ann Neurol. 2017 May;81(5):641-652. doi: 10.1002/ana.24922. Epub 2017 May 4. PMID 28318037
- [Result] Garone C, Garcia-Diaz B, Emmanuele V, Lopez LC, Tadesse S, Akman HO, Tanji K, Quinzii CM, Hirano M. Deoxypyrimidine monophosphate bypass therapy for thymidine kinase 2 deficiency. EMBO Mol Med. 2014 Aug;6(8):1016-27. doi: 10.15252/emmm.201404092. PMID 24968719
- [Result] Chanprasert S, Wang J, Weng SW, Enns GM, Boue DR, Wong BL, Mendell JR, Perry DA, Sahenk Z, Craigen WJ, Alcala FJ, Pascual JM, Melancon S, Zhang VW, Scaglia F, Wong LJ. Molecular and clinical characterization of the myopathic form of mitochondrial DNA depletion syndrome caused by mutations in the thymidine kinase (TK2) gene. Mol Genet Metab. 2013 Sep-Oct;110(1-2):153-61. doi: 10.1016/j.ymgme.2013.07.009. Epub 2013 Jul 17. PMID 23932787